CLINICAL TRIAL: NCT00678457
Title: Ondansetron With Olanzapine for the Treatment of Alcohol Dependence: A Preliminary Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Bankole Johnson, DSc, M.D., Ph.D., University of Virginia
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TO45228; IRB-HSR #12816
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; alcohol abuse; drinking; alcohol
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ondansetron/olanzapine (Experimental): ondansetron (4 μg/kg b.i.d.)
  olanzapine (9 μg/kg)
  Interventions: Drug: Ondansetron; Drug: Olanzapine
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — ondansetron (4 μg/kg b.i.d.)
  Other Names: Zofran
  Arms: ondansetron/olanzapine
Drug: Olanzapine — olanzapine (9, 18, and 36 μg/kg)
  Other Names: Zyprexa
  Arms: ondansetron/olanzapine
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
This study would like to test whether the combination of ondansetron and olanzapine will be superior to placebo at decreasing self-reported heavy drinking among early onset alcoholics.

DETAILED DESCRIPTION:
Target population: We will enroll male and female who meet DSM IV criteria for alcohol dependence and who are currently drinking equal or more than 21 alcohol units/week for women and equal or more than 28 alcohol units/week for men in the 7 day period prior to enrollment.

This is a double-blind placebo-controlled study. Eligible subjects will be randomized to ondansetron (4 ug/kg) and olanzapine (9, 18, 36 ug/kg) vs placebo. All subjects will participate in a 9 week regimen of weekly BBCET and outpatient medication treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* Aged 18 years and above and weighing ≥40 kg and ≤140 kg
* Drinking on average ≥21 and ≥28 drinks/week for women and men, respectively, in the 7-day period prior to enrollment
* DSM-IV-R diagnosis of alcohol dependence
* Good physical health as determined by a complete physical examination, electrocardiogram (EKG) within normal limits and laboratory screening tests within acceptable range
* Negative pregnancy test at intake.
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments
* Willing to participate in behavioral treatments for alcoholism
* Answer an advertisement in the newspaper/radio/television, and express a wish to stop drinking
* Provide evidence of stable residence in the last month prior to enrollment in the study, and have no plans to move in the next three months

Exclusion Criteria:

* Any current axis I DSM-IV psychiatric disorder other than alcohol or nicotine dependence that warrants treatment or would preclude safe participation in the protocol
* Severe alcohol withdrawal symptoms that, in the physician's opinion, require inpatient treatment
* Serious medical comorbidity requiring medical intervention or close supervision, or any condition that can interfere with the receipt of ondansetron or olanzapine
* Severe or life-threatening adverse reactions to the ondansetron or olanzapine medications in the past or during this clinical trial
* Female subjects who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study
* Received inpatient or outpatient treatment for alcohol dependence within the last 30 days
* Significant medical illness (including hypertension) as determined by history and/or complete physical examination.
* Gross neurological disease
* Mental retardation
* Pyrexia of unknown origin
* Diagnosis or suspicion of Alzheimer's disease
* Clinically significant abnormalities on the EKG that will preclude safe participation
* Recent (last 3 months) history of ischemic heart disease or myocardial infarction.
* Current infective hepatitis as evidenced by clinical manifestations. If hepatitis is suspected, a hepatitis antibody/antigen screen will be done.
* Participation in a clinical study within the last 30 days
* Elevation of liver enzymes
* History of any severe or life-threatening reaction to olanzapine or ondansetron
* Past or current history of seizures disorder
* Past or current history of diabetes
* Being treated with any medication with potential for clinically significant interactions with alcohol or olanzapine and/or ondansetron. These include:, serotonin antagonists (e.g., ritanserin or buspirone), dopamine antagonists (e.g., haloperidol), or compounds with actions similar to disulfiram (Antabuse®).
* Pending imprisonment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The combination of ondansetron and olanzapine will be safe and superior to placebo at decreasing self-reported heavy drinking among early-onset alcoholics. | Throughout the study

SECONDARY OUTCOMES:
The combination of ondansetron and olanzapine will be superior to placebo at reducing the psychosocial consequences of drinking. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc, MD, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia